CLINICAL TRIAL: NCT05884164
Title: Comparative Study: Erector Spinae Plane Block Versus Paravertebral Plane Block Regarding Their Effect on Peri-operative Opioid Consumption in Patients Undergoing Minimally Invasive Mitral Valve Replacement .
Brief Title: ESPB Versus PVPB Regarding Their Effect on Peri-operative Opioid Consumption in Patients Undergoing Minimally Invasive Mitral Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FMASU MD89 / 2022
Record Dates: First submitted 2023-04-01; First posted 2023-06-01 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: ERAS; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae group (Active Comparator): Patients will receive erector spinae plane block after general anaesthesia .
  Interventions: Procedure: Thoracic erector spinae plane block
- Paravertebral block group (Active Comparator): Patients will receive paravertebral plane block after general anaesthesia .
  Interventions: Procedure: Thoracic paravertebral plane block

INTERVENTIONS:
Procedure: Thoracic erector spinae plane block — After induction of general Anaesthesia,a high frequency ultrasound probe will be placed in a longitudinal orientation 3 cm from the midline. Once the erector spinal muscle and the transverse processes are identified, spinal needle will be inserted after standard skin disinfection in a caudal to cephalad direction using a sterile probe cover until the tip lay in the interfacial plane deep to the erector spinal muscle. After hydrolocalization with ml normal saline, this plane will be opened and 20 ml of 0.25 %bupivacaine will be administered for block performance
  Arms: Erector spinae group
Procedure: Thoracic paravertebral plane block — After induction of general Anaesthesia ,with the probe in the longitudinal paramedian position, it is then moved from medial to lateral direction to appreciate the saw tooth appearance of the facet joints close to the midline which changes to long finger-like shadow of the transverse process as the probe is moved slightly laterally. Repositioning the probe over the transverse process ensuring the space of interest is in the middle of the probe once again one should appreciate the intercostal muscles and the dense bright white line of the pleura in between the shadows of the transverse processes. The needle is then introduced at the caudal end of the probe in plane in a caudal to cranial direction aiming for the angle between the bottom of the transverse process and the pleura. Once position is confirmed, 20 ml of 0.25% bupivacaine will be administered for the block performance.
  Arms: Paravertebral block group

SUMMARY:
In recent years , the popularity of ultrasound-guided fascial plane blocks has increased in achieving an effective postoperative analgesia and hence achieving enhanced recovery after surgery (ERAS) .

Mastering the use of ultrasound encourages anesthetists on the frequent use of regional anesthesia . Fascial plane blocks are increasingly becoming a part of multimodal analgesia as an alternative pain management strategy in cardiac surgery. Various regional techniques especially paravertebral plane blocks have been recently described to reduce the postoperative pain in cardiac surgery with enhanced recovery . Ultrasound-guided erector spinae plane block is a recently introduced technique for regional analgesia in thoracic neuropathic pain, rib fractures, and breast surgeries. This study aims to compare between the two techniques regarding their peri-operative analgesic effect and their impact on enhanced recovery after surgery.

DETAILED DESCRIPTION:
This study aims to compare between the effectiveness of Erector spinae plane block and thoracic paravertebral plane block in reducing the perioperative need of opioids in patients undergoing minimally invasive mitral valve replacement as part of ERAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) score III.
* Patients aged ≥ 18 years old.
* Patients scheduled for minimally invasive mitral valve replacement through a right mini thoracotomy.

Exclusion Criteria:

* Patients refusing to be involved in this study.
* Patients with ASA score > III.
* Patients aged < 18 years.
* Patients with local infection at the site of needle puncture.
* Patients with known hypersensitivity to local anesthetic (LA).
* Patients with hepatic or renal impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
intraoperative opioid consumption | Through intraoperative period, average of 6 hours
  Fentanyl in micrograms intraoperatively
Postoperative opioid consumption | For 24 hours after extubation
  morphine in milligram postoperatively

SECONDARY OUTCOMES:
Time for extubation | 24 hours postoperative
  The time it took for the patient to be extubated in ICU
Time for ambulation | Through the stay of the patient in ICU postoperatively, average of 2 days.
  The time when the patient is ambulated in the ICU
Postoperative respiratory depression | 24 hours after extubation
  Determined by respiratory rate
Postoperative respiratory depression | 24 hours after extubation
  Determined by oxygen saturation
Postoperative respiratory depression | 24 hours after extubation
  Determined by the need of oxygen support after extubation
Length of ICU stay | Through patient's stay inicu till discharge to ward, average of 3 days
  The time patient spends in the ICU postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Galal A El Kadi, MD, Study Chair — Ain Shams University; Mohamed S Zaki, MD, Study Chair — Ain Shams University; Mona M Ammar, MD, Study Chair — Ain Shams University; Islam A Abdelmouty, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: No